CLINICAL TRIAL: NCT06023485
Title: The Effect of Stress Ball Use on Procedural Pain Caused by Subcutaneous Injection in Orthopedic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Figen Dıgın, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: The Effect of Stress Ball Use; KLÜBAP-249 (Other Grant/Funding Number: KLÜBAP-249); 2023-249 (Other Grant/Funding Number: 2023-249); 2023-249 (Other: Kırklareli university)
Record Dates: First submitted 2023-08-27; First posted 2023-09-05 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Misadventure During Injection / Vaccination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (stress ball) (Experimental): The patients in the experimental group will be given a stress ball before the SC injection during the routine daytime treatment of the ward at 10:00. The patient will be asked to squeeze the stress ball with his hand on the opposite extremity of the upper extremity where SC injection was applied, counting to five, and then to relax his hand. In the meantime, 0.4 ml of LMWH will be administered by SC route according to the doctor's request. During the patient's drug administration and 2 minutes after the application. The level of pain in the area where SC was applied will be evaluated with VAS.
  Interventions: Other: stress ball use during subcutaneous injection
- Control group (No Intervention): For the patients in the control group, 0.4 ml of LMWH will be administered by the nurse in the routine daytime treatment of the service at 10:00, according to the doctor's request. During the patient's drug administration and 2 minutes after the application. The level of pain in the area where SC was applied will be evaluated with VAS.

INTERVENTIONS:
Other: stress ball use during subcutaneous injection — The effect of stress ball use on pain during subcutaneous injection
  Arms: Experimental group (stress ball)

SUMMARY:
Randomization in the study will be done by the researchers with the Randomizer Research program. The research will be carried out between 01.01.2023 and 01.10.2023 with the participation of 134 patients who were hospitalized in the postoperative period at Trakya University Health Research and Application Center Orthopedics and Traumatology Service and participated voluntarily. In the study, in the G.Power 3.1.9.4 program, the effect size was 0.5, the confidence level was 95%, and the power was 80%, and the minimum sample size to be reached was 134 patients (67 experiments- 67 controls), each group consisting of 67 people. Before the study, all patients will be informed by the researchers, and written consent will be obtained from the patients who volunteered to participate in the study. All patients will be asked the questions in the Patient Information Form and the pretest Vizuel Analog Scala (VAS) scores in the Patient follow-up form will be recorded before the subcutaneous (SC) injection application. The patients in the experimental group will be given a stress ball before the SC injection during the routine daytime treatment of the ward at 10:00. The patient will be asked to squeeze the stress ball with his hand on the opposite extremity of the upper extremity where SC injection was applied, counting to five, and then to relax his hand. The level of pain in the area where SC was applied will be evaluated with VAS. For the patients in the control group, 0.4 ml of LMWH will be administered by the nurse in the routine daytime treatment of the service at 10:00, according to the doctor's request. During the patient's drug administration and 2 minutes after the application. The level of pain in the area where SC was applied will be evaluated with VAS.

DETAILED DESCRIPTION:
The ramdomized research will be carried out between 01.01.2023 and 01.10.2023 with the participation of 134 patients who were hospitalized in the postoperative period at Trakya University Health Research and Application Center Orthopedics and Traumatology Service and participated voluntarily. In the study, in the G.Power 3.1.9.4 program, the effect size was 0.5, the confidence level was 95%, and the power was 80%, and the minimum sample size to be reached was 134 patients (67 experiments- 67 controls), each group consisting of 67 people. The study included 18 patients who were hospitalized in the orthopedics and traumatology clinic, were in the post-operative period, were not diabetic, conscious, cooperative and oriented (without delirium, etc.), without a diagnosis of psychiatric disease, who could localize the pain, did not undergo upper extremity surgery, and volunteered to participate in the study. Age and older patients will be included. Before the study, all patients will be informed by the researchers, and written consent will be obtained from the patients who volunteered to participate in the study. All patients will be asked the questions in the Patient Information Form and the pretest Vizuel Analog Scala (VAS) scores in the Patient follow-up form will be recorded before the subcutaneous (SC) injection application. The patients in the experimental group will be given a stress ball before the SC injection during the routine daytime treatment of the ward at 10:00. The patient will be asked to squeeze the stress ball with his hand on the opposite extremity of the upper extremity where SC injection was applied, counting to five, and then to relax his hand. In the meantime, 0.4 ml of LMWH will be administered by SC route according to the doctor's request. During the patient's drug administration and 2 minutes after the application. The level of pain in the area where SC was applied will be evaluated with VAS. For the patients in the control group, 0.4 ml of LMWH will be administered by the nurse in the routine daytime treatment of the service at 10:00, according to the doctor's request. During the patient's drug administration and 2 minutes after the application. The level of pain in the area where SC was applied will be evaluated with VAS. Unlike the control group, the patients in the experimental group will be asked to tighten and loosen the stress ball during SC injection

ELIGIBILITY:
Inclusion Criteria:

* patients;
* who were hospitalized in the orthopedics and traumatology clinic,
* who were in the post-operative period,
* who were not diabetic,
* who were conscious,
* who were cooperative and oriented (without delirium, etc.),
* who were not diagnosed with psychiatric disease,
* who could localize pain,
* who did not undergo upper extremity surgery, and
* who volunteered to participate in the study.

Exclusion Criteria:

* Patients who do not volunteer to participate in the study will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
pain management during subcutaneous injection | 9 months
  The patient will be asked to squeeze the stress ball with his hand on the opposite extremity of the upper extremity where SC injection was applied, counting to five, and then to relax his hand. In the meantime, 0.4 ml of LMWH will be administered by SC route according to the doctor's request. During the patient's drug administration and 2 minutes after the application. The level of pain in the area where SC was applied will be evaluated with Vizuel Analog Scala (VAS). The VAS is a unidimensional scale frequently used to measure pain severity. The scale consists of a 10-cm demarcated line in which 0 cm represents no pain and 10 cm represents unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No